CLINICAL TRIAL: NCT04468373
Title: Study of the WA-NG (NG-IMT) Telescope Prosthesis in Patients With Central Vision Impairment Associated With End-Stage Age Related Macular Degeneration
Brief Title: Study of WA-NG (NG-IMT) Telescope Prosthesis in Patients With End-stage Age-related Macular Degeneration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Development of next-generation device
Sponsor: VisionCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA-NG-001 EUROPE
Record Dates: First submitted 2018-12-13; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2018-12

CONDITIONS: Age Related Macular Degeneration
Keywords: Macular Degeneration; Visual Impairment; Implantable Telescope
MeSH Terms: conditions — Macular Degeneration; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WA-NG (NG-IMT) Telescope Prothesis (Experimental): Implantable Miniature Telescope for end stage AMD (Age-related Macular Degeneration)
  Interventions: Device: WA-NG (NG-IMT) Telescope Prothesis

INTERVENTIONS:
Device: WA-NG (NG-IMT) Telescope Prothesis — The WA-NG telescope prosthesis is the next generation telescopic implantable device which, when combined with the optics of the cornea, constitutes a telephoto system for improvement of visual acuity in patients with severe to profound vision impairment due to bilateral, end-stage age-related macular degeneration. The device is implanted in one of the patient's eyes. In this way, the implanted eye provides central vision and the non-implanted eye can continue to provide peripheral vision.

SUMMARY:
The purpose of this study is to evaluate the safety of the updated Model WA-NG telescope prosthesis (hereafter WA-NG telescope), an injectable telescope device, in patients with bilateral moderate to profound central vision impairment due to end-stage age-related macular degeneration.

DETAILED DESCRIPTION:
Patients will be screened for eligibility and informed consent will be obtained from those who meet screening criteria and are interested in participating in the study. Eligible patients will be examined preoperatively to obtain a medical history and to establish a baseline for ocular condition.

Postoperatively, patients will undergo ophthalmic evaluation at regular intervals as specified in this protocol.

ELIGIBILITY:
**The following Inc. & Exc. are sample and not completed list **

Main Exclusion Criteria:

* Patients with bilateral, stable, moderate to profound central vision impairment due to bilateral central scotoma associated with end-stage macular degeneration, defined as retinal findings of bilateral, geographic atrophy or disciform scar with foveal involvement.
* Patients must have distance BCVA between 20/80 and 20/800, and adequate peripheral vision in one eye (the non-implanted eye) to allow navigation
* Patients must achieve at least a five letter improvement on the ETDRS chart in the eye scheduled for surgery, with the external telescope simulator (ETS)
* Patients must be available for the study duration of 12 months
* Patients must be alert, mentally competent, and able to understand and comply with the requirements of the clinical trial, and be personally motivated to abide by the requirements and restrictions of the clinical trial.

Main Exclusion Criteria:

* Evidence of active CNV on fluorescein angiography or treatment for CNV within the past six months.
* Patients who may require fellow eye cataract extraction and intraocular lens implantation during the 12 months following WA-NG telescope implantation. If fellow eye cataract extraction is anticipated, this procedure should be performed at least 30 days prior to enrollment in the clinical study.
* Patients who have had or are expected to have ophthalmic related surgery within the 30 days preceding implantation of the device.
* Patients who have undergone previous intraocular or corneal surgery of any kind in the operative eye(s), including any type of surgery for either refractive or therapeutic purposes.
* Patients participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Positional stabilitytilt (the following parameter will be measured/ assessed :device centered (yes/ no) questionnaire) | 12 months
  Device positional stability will be assessed by slit lamp examination (microscope with a bright light used during an eye exam) and anterior segment Ocular Coherence Tomography (OCT is a non-invasive imaging test )
Positional stabilitytilt, the following parameter will be measured/ assessed : tilted (° C) | 12 months
  Device positional stability will be assessed by slit lamp examination (microscope with a bright light used during an eye exam) and anterior segment Ocular Coherence Tomography (OCT is a non-invasive imaging test )
Positional stabilitytilt , the following parameter will be measured/ assessed : malpositioned (yes/no) questionnaire | 12 months
  Device positional stability will be assessed by slit lamp examination (microscope with a bright light used during an eye exam) and anterior segment Ocular Coherence Tomography (OCT is a non-invasive imaging test )
Positional stabilitytilt , the following parameter will be measured/ assessed : endothelial cell count (Cells/mm2)) | 12 months
Positional stabilitytilt , the following parameter will be measured/ assessed : Intraocular pressure (mmHg) | 12 months
  Device positional stability will be assessed by slit lamp examination (microscope with a bright light used during an eye exam)
Number of Adverse events associated with the implant and use of the device will be evaluated. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Diane Gordon, Study Director — VisionCare Ophthalmic Technologies
Locations (2):
- Mater Private Hospital, Dublin, Ireland
- VISSUM Ophthalmological Corporation, Alicante, Spain